CLINICAL TRIAL: NCT04708444
Title: Prognostic Value of CD318 in Acute Myeloid Leukemia Patients at Assiut University Hospital
Brief Title: Prognostic Value of CD318 in AML at Assiut University Hospital.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shimaa Arafa Ibrahim (Other)
Responsible Party: Sponsor-Investigator, Shimaa Arafa Ibrahim, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: CD318 in AML
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: CD318 — Flowcytometric marker

SUMMARY:
We will focus on the prognostic value of CD318 in acute myeloid leukemia patients at Assiut University Hospital

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a disease with high mortality and variable prognosis . It remains a disease with a highly variable outcome depending on the exact footprint of the AML .Although many patients with AML have a response to induction therapy ,refractory disease is common and relapse represents the major cause of treatment failure .In 2016 the World Heath Organization published revisions to classification of Myeloid Neoplasms and Acute leukemias .Well-established prognostic factors are cytogenetic aberrations such as t(8;21), inv(16), and t(15;17) as well as mutated IDH1/2, NPM1, and FLT3 genes but only few markers can specifically predict the outcome after HSCT .Immunophenotyping via flowcytometry comprises an additional fast technique to predict outcome in AML, although only few markers are yet established as prognostic factors in clinical routine diagnosis, despite the fact that new and rapidly available markers are needed to improve the treatment decisions in AML patients. This is even more since starting therapy in AML patients must be initiated immediately after diagnosis . Overall mortality from AML is high and treatment should be initiated within hours after first diagnosis . In hematopoietic cells,CD318 has been identified as stem cell marker for both benign and malignant progenitor cells. CD318+ bone marrow or cord blood-derived cells have been shown to be capable to initiate multi-lineage hematopoiesis in vitro and in vivo .CD318 (CUB domain containing protein-1, CDCP1) is a highly glycosylated single pass transmembrane protein express endomesenchymal and neural stem cells and fibroblasts and hematopoietic.Overexpression of CD318 has been recently correlated with poor overall survival(OS) in colonic ,breast ,renal, hepatocellular ,and pancreatic Carcinoma.possibly due to its role in metastasis formation via interaction with integrins and anti-apoptotic signaling via Akt. Of AML blasts, pronounced CD318 expression has been observed on the immature CD34+CD133+ leukemic cells subset implicated to be enriched for leukemic stem. However, the impact of CD318 on survival in hematological malignancies has so far not been analyzed. Study done by Jonas S et al showed 57% of AML patients expressed relevant CD318 levels and a significant correlation of CD 318 surface levels with prognosis was observed . In our study investigators will use flowcytometry to detect CD318 on AML blasts and correlate it with disease course and outcome.

ELIGIBILITY:
Inclusion Criteria:

1. newly diagnosed AML patients
2. Age more than 18 years
3. Patients not starting chemotherapy yet
4. Primary AML
5. Secondary AML on top of MDS or myeloproliverative noeplasms

Exclusion Criteria:

1. Refractory AML patients
2. Relapsed AML patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: our study will include newly diagnosed AML patients at clinical hematology unit Assiut University during the period from March 2021 to August 2022. The diagnosis and classification of AML relied on morphology and cytochemistry of bone marrow according to FAB classification. patients will be subjected to full history taking clinical examination laboratory investigations CBC,LFTs,RFTs,electrolytes,ESR,LDH,CRP,Coagulationprofile,aptt ,fibrinogen, D dimer, bone marrow assessment with immunephenotyping and cytogenetic analysis.
  Flowcytometric analysis of AML blasts for CD 318
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Prognosis of CD318 in AML | Throughout study completion, average of one year
  Flowcytometric analysis of AML blasts for CD318 and correlate it with disease course (progression free survival) and disease outcome (overall survival) . Also correlate level of expression of CD318 with response to treatment given ( intensive chemotherapy, hypomethylating agents, alternative palliative therapy.
  CD318 to detect level of expression and correlate it with disease course (progression free survival) and outcome (overall survival) .

REFERENCES:
- [Background] Grimwade D, Walker H, Oliver F, Wheatley K, Harrison C, Harrison G, Rees J, Hann I, Stevens R, Burnett A, Goldstone A. The importance of diagnostic cytogenetics on outcome in AML: analysis of 1,612 patients entered into the MRC AML 10 trial. The Medical Research Council Adult and Children's Leukaemia Working Parties. Blood. 1998 Oct 1;92(7):2322-33. PMID 9746770
- [Background] Grimwade D, Walker H, Harrison G, Oliver F, Chatters S, Harrison CJ, Wheatley K, Burnett AK, Goldstone AH; Medical Research Council Adult Leukemia Working Party. The predictive value of hierarchical cytogenetic classification in older adults with acute myeloid leukemia (AML): analysis of 1065 patients entered into the United Kingdom Medical Research Council AML11 trial. Blood. 2001 Sep 1;98(5):1312-20. doi: 10.1182/blood.v98.5.1312. PMID 11520776
- [Background] Kottaridis PD, Gale RE, Frew ME, Harrison G, Langabeer SE, Belton AA, Walker H, Wheatley K, Bowen DT, Burnett AK, Goldstone AH, Linch DC. The presence of a FLT3 internal tandem duplication in patients with acute myeloid leukemia (AML) adds important prognostic information to cytogenetic risk group and response to the first cycle of chemotherapy: analysis of 854 patients from the United Kingdom Medical Research Council AML 10 and 12 trials. Blood. 2001 Sep 15;98(6):1752-9. doi: 10.1182/blood.v98.6.1752. PMID 11535508
- [Background] Conze T, Lammers R, Kuci S, Scherl-Mostageer M, Schweifer N, Kanz L, Buhring HJ. CDCP1 is a novel marker for hematopoietic stem cells. Ann N Y Acad Sci. 2003 May;996:222-6. doi: 10.1111/j.1749-6632.2003.tb03249.x. PMID 12799299
- [Background] Scherl-Mostageer M, Sommergruber W, Abseher R, Hauptmann R, Ambros P, Schweifer N. Identification of a novel gene, CDCP1, overexpressed in human colorectal cancer. Oncogene. 2001 Jul 19;20(32):4402-8. doi: 10.1038/sj.onc.1204566. PMID 11466621
- [Background] Hooper JD, Zijlstra A, Aimes RT, Liang H, Claassen GF, Tarin D, Testa JE, Quigley JP. Subtractive immunization using highly metastatic human tumor cells identifies SIMA135/CDCP1, a 135 kDa cell surface phosphorylated glycoprotein antigen. Oncogene. 2003 Mar 27;22(12):1783-94. doi: 10.1038/sj.onc.1206220. PMID 12660814
- [Background] Casar B, Rimann I, Kato H, Shattil SJ, Quigley JP, Deryugina EI. In vivo cleaved CDCP1 promotes early tumor dissemination via complexing with activated beta1 integrin and induction of FAK/PI3K/Akt motility signaling. Oncogene. 2014 Jan 9;33(2):255-68. doi: 10.1038/onc.2012.547. Epub 2012 Dec 3. PMID 23208492
- [Background] Liersch R, Muller-Tidow C, Berdel WE, Krug U. Prognostic factors for acute myeloid leukaemia in adults--biological significance and clinical use. Br J Haematol. 2014 Apr;165(1):17-38. doi: 10.1111/bjh.12750. Epub 2014 Feb 1. PMID 24484469
- [Background] Uekita T, Fujii S, Miyazawa Y, Iwakawa R, Narisawa-Saito M, Nakashima K, Tsuta K, Tsuda H, Kiyono T, Yokota J, Sakai R. Oncogenic Ras/ERK signaling activates CDCP1 to promote tumor invasion and metastasis. Mol Cancer Res. 2014 Oct;12(10):1449-59. doi: 10.1158/1541-7786.MCR-13-0587. Epub 2014 Jun 17. PMID 24939643
- [Background] Alajati A, Guccini I, Pinton S, Garcia-Escudero R, Bernasocchi T, Sarti M, Montani E, Rinaldi A, Montemurro F, Catapano C, Bertoni F, Alimonti A. Interaction of CDCP1 with HER2 enhances HER2-driven tumorigenesis and promotes trastuzumab resistance in breast cancer. Cell Rep. 2015 Apr 28;11(4):564-76. doi: 10.1016/j.celrep.2015.03.044. Epub 2015 Apr 16. PMID 25892239
- [Background] Dohner H, Weisdorf DJ, Bloomfield CD. Acute Myeloid Leukemia. N Engl J Med. 2015 Sep 17;373(12):1136-52. doi: 10.1056/NEJMra1406184. No abstract available. PMID 26376137
- [Background] Schmid C, Labopin M, Socie G, Daguindau E, Volin L, Huynh A, Bourhis JH, Milpied N, Cornelissen J, Chevallier P, Maertens J, Jindra P, Blaise D, Lenhoff S, Ifrah N, Baron F, Ciceri F, Gorin C, Savani B, Giebel S, Polge E, Esteve J, Nagler A, Mohty M; Acute Leukemia Working Party of the European Group of Blood and Bone Marrow Transplantation. Outcome of patients with distinct molecular genotypes and cytogenetically normal AML after allogeneic transplantation. Blood. 2015 Oct 22;126(17):2062-9. doi: 10.1182/blood-2015-06-651562. Epub 2015 Sep 8. PMID 26351297
- [Background] Arber DA, Orazi A, Hasserjian R, Thiele J, Borowitz MJ, Le Beau MM, Bloomfield CD, Cazzola M, Vardiman JW. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016 May 19;127(20):2391-405. doi: 10.1182/blood-2016-03-643544. Epub 2016 Apr 11. PMID 27069254
- [Background] De Kouchkovsky I, Abdul-Hay M. 'Acute myeloid leukemia: a comprehensive review and 2016 update'. Blood Cancer J. 2016 Jul 1;6(7):e441. doi: 10.1038/bcj.2016.50. PMID 27367478
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Enyindah-Asonye G, Li Y, Ruth JH, Spassov DS, Hebron KE, Zijlstra A, Moasser MM, Wang B, Singer NG, Cui H, Ohara RA, Rasmussen SM, Fox DA, Lin F. CD318 is a ligand for CD6. Proc Natl Acad Sci U S A. 2017 Aug 15;114(33):E6912-E6921. doi: 10.1073/pnas.1704008114. Epub 2017 Jul 31. PMID 28760953
- [Background] Estey EH. Acute myeloid leukemia: 2019 update on risk-stratification and management. Am J Hematol. 2018 Oct;93(10):1267-1291. doi: 10.1002/ajh.25214. PMID 30328165
- [Background] Heitmann JS, Hagelstein I, Hinterleitner C, Roerden M, Jung G, Salih HR, Marklin M, Kauer J. Identification of CD318 (CDCP1) as novel prognostic marker in AML. Ann Hematol. 2020 Mar;99(3):477-486. doi: 10.1007/s00277-020-03907-9. Epub 2020 Jan 21. PMID 31965270